CLINICAL TRIAL: NCT05653115
Title: Outcomes of Bariatric Surgery in the Setting of Compensated Advance+B9d Chronic Liver Disease Associated With Clinically Significant Portal Hypertension
Brief Title: Portal Hypetension and Bariatric Surgery (BARIAPORTAL)
Acronym: BARIAPORTAL
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 22Chirdig01
Record Dates: First submitted 2022-11-15; First posted 2022-12-16 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Bariatric Surgery Candidate; Obesity, Morbid; Portal Hypertension
MeSH Terms: conditions — Obesity, Morbid; Hypertension, Portal | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Bariatric surgery: Individuals with morbid obesity and clinically relevant portal hypertension undergoing bariatric surgery
  Interventions: Procedure: Bariatric surgery

INTERVENTIONS:
Procedure: Bariatric surgery — Bariatric surgery

SUMMARY:
The worldwide obesity epidemic has led to an increase in the proportion of patients with chronic liver disease due to non-alcoholic fatty liver disease (NAFLD) and in the prevalence of obesity in patients with cirrhosis of all etiologies. The reported prevalence of obesity in patients with cirrhosis is of 30% which appears similar to that of the general population.

Bariatric surgery is currently considered as the most effective and durable means for the management of morbid obesity as it is associated with the remission and/or improvement of many obesity associated comorbidities as well as improved quality and expectancy of life.

However, the surgical risk is increased compared to individuals without cirrhosis, and determining the risk/benefit ratio of bariatric surgery in the setting of cirrhosis is a complex task further hampered by the lack of randomized controlled trials.

The Nationwide Inpatient Sample study reported a slightly increased rate of mortality of bariatric surgery in the setting of compensated cirrhosis compared to individuals without cirrhosis (0.9% vs 0.3%). Interestingly, this risk was as high as 16.3% in individuals with decompensated cirrhosis (16.3%). However, this study has been published more than 10 years ago and the mortality of bariatric surgery has decreased significantly and is around 0.1%. Furthermore, the introduction of transient elastography in clinical practice has allowed the early identification of patients with chronic liver disease (CLD) at risk of developing clinically significant portal hypertension (CSPH).

A few series including a limited number of patients have been published indicating that CSPH should not be considered as a formal contraindication for bariatric surgery.

This study is meant to assess the outcomes of bariatric surgery in patients with morbid obesity and compensated advanced chronic liver disease (cACLD) (currently synonymous of the term "compensated cirrhosis'') associated with clinically significant portal hypertension (CSPH) in a large multicentric, multinational series.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with morbid obesity (BMI > 40 or 35 with at least one comorbidity) undergoing bariatric surgery and CSPH (defined as HVPG > 10 mmHg and/or cross-sectional imaging showing collateral circulation, and/or varices at esophagogastroduodenoscopy.
* Information available to determine postoperative mortality (at least first postoperative month of any duration in case of primary hospitalization longer than 1 month)

Exclusion Criteria:

* Absence of preoperative evidence of CSPH in spite of evidence liver cirrhosis.
* Absence of information to determine at least postoperative mortality.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with morbid obesity and clinically relevant portal hypertension undergoing bariatric surgery
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2022-01-12 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Postoperative mortality | Within 90 of surgery or any tipe during postoperative hospital stay
  number of patients who died after the surgery

SECONDARY OUTCOMES:
General information and anthropometrics | through study completion on average 1 year
  Age (years), gender (male/ female), body weight (Kg), height (meters), BMI (body weight in Kg/height in meters); obesity linked comorbid conditions : hypertension (HT is defined as resting blood pressure persistently ≥ 140/90 mmHg or need for antihypertensive drugs), Type 2 diabetes (T2D is defined as fasting glucose > 7.0 mmol/L after two measurements or need for oral antidiabetics), sleep apnea syndrome (SAS is quantified by sleep studies).
Etiology of liver cirrhosis | through study completion on average 1 year
  viral (HCV, HBV), NASH, Alcohol, other
Preoperative work-up to define CSPH | through study completion on average 1 year
  endoscopy (presence of varices), imaging CT scan (presence of porto-systemic shunts), MRI (presence of porto-systemic shunts), portal pressure measure (mmHg).
Liver function | through study completion on average 1 year
  Child's score (Child A 5-6 points; Child B 7-9; Child C 10-15), Model for End-Stage Liver Disease (MELD) score (number of points up to 40)
Strategy to lower portal hypertension | through study completion on average 1 year
  TIPS, Beta blockers
Type of bariatric procedure | through study completion on average 1 year
  SG, RYGB, Band, other
Postoperative complications | through study completion on average 1 year
  bleeding, leak, pulmonary embolus, stricture, other
Functional results | through study completion on average 1 year
  weight loss in Kg as compared to preoperative weight

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de NICE, Nice, France

IPD SHARING:
Plan to Share IPD: No
Not scheduled

REFERENCES:
- [Background] Temime V, Ghanem OM, Heimbach JK, Diwan TS, Tranchart H, Abdallah H, Blanchard C, Lontrichard M, Reche F, Borel AL, Belluzzi A, Foletto M, Manno E, Poghosyan T, Chierici A, Iannelli A. Outcomes of bariatric surgery in the setting of compensated advanced chronic liver disease associated with clinically significant portal hypertension: a multicenter, retrospective, cohort study on feasibility and safety. Int J Surg. 2024 Jun 1;110(6):3562-3570. doi: 10.1097/JS9.0000000000001310. PMID 38819255